CLINICAL TRIAL: NCT00651547
Title: A 12 Week Randomized, Double-Blind, Double-Dummy, Placebo-Controlled Trial of Symbicort TM (40/4.5 Mcg) Versus Its Mono-Products (Budesonide and Formoterol) in Asthmatic Children Aged Six to Eleven Years - SEEDLING 40/4.5
Brief Title: Symbicort in Asthmatic Children - SEEDLING
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SD-039-0718; D5896C00718
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: Asthma; Symbicort; budesonide/formoterol; budesonide; formoterol; children
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: budesonide/formoterol
- 2 (Active Comparator)
  Interventions: Drug: budesonide
- 3 (Active Comparator)
  Interventions: Drug: formoterol

INTERVENTIONS:
Drug: budesonide/formoterol
  Other Names: Symbicort
  Arms: 1
Drug: budesonide
  Arms: 2
Drug: formoterol
  Arms: 3

SUMMARY:
The purpose of this study is to compare Symbicort with budesonide alone and formoterol alone in the treatment of asthma in children aged 6 to 11 years

ELIGIBILITY:
Inclusion Criteria:

* Baseline lung function tests results as determined by the protocol
* Required and received treatment with inhaled corticosteroids within the timeframe and doses specified in the protocol

Exclusion Criteria:

* Has required treatment with non-inhaled corticosteroids within previous 4 weeks, has sensitivity to drugs specified in the protocol or requires treatment with beta-blockers
* Has been hospitalised or required emergency treatment for asthma-related condition within previous 6 months
* Has had cancer within previous 5 years or has a significant disease, as judged by investigator, that may put the patient at risk in this study

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 405 (Estimated)
Dates: Start 2002-07; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Morning PEF | Daily

SECONDARY OUTCOMES:
Lung function, asthma symptoms, use of rescue medication, adverse events and other safety assessments | Throughout the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bonuccelli, Study Director — AstraZeneca